CLINICAL TRIAL: NCT00409097
Title: Effect of Rosiglitazone on ADMA in Critical Illness
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Amsterdam UMC, location VUmc (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HK0506
Record Dates: First submitted 2006-12-07; First posted 2006-12-08 (Estimated); Last update posted 2006-12-08 (Estimated); Status verified 2006-12

CONDITIONS: Critical Illness; Multiple Organ Failure
Keywords: ADMA; MOF; Critical illness
MeSH Terms: conditions — Critical Illness; Multiple Organ Failure | interventions — Rosiglitazone

INTERVENTIONS:
Drug: Rosiglitazone

SUMMARY:
The purpose of this study is to determine whether Rosiglitazone,decreases the ADMA concentration and thereby increases the arginine/ADMA ratio of critically ill patients.

DETAILED DESCRIPTION:
Endothelial vasodilatation dysfunction precedes the development of arteriosclerosis. The endothelium plays a pivotal role in the control of the vascular tone by releasing nitric oxide (NO). The amino acid arginine is the sole substrate for the enzyme NO synthase (NOS). Asymmetric dimethylarginine (ADMA) is an endogenous derivative of arginine that inhibits NOS. Thus the arginine/ADMA ratio an important determinant of NO production by NOS. ADMA is an independent risk factor for cardiovascular disease, but elevated levels of ADMA have also been shown to be a strong independent predictor of ICU mortality. The central mechanism by which ADMA may cause deterioration in critically ill patients is by impairing organ blood flow and reducing cardiac function, especially during stress. Accumulation of ADMA could thereby be a causative factor in the development multi organ failure (MOF). Thus inhibition of NO production by ADMA may become especially important when cardiac demand is increased.

ELIGIBILITY:
Inclusion Criteria:

* critically ill patients
* age between 18 and 75 years
* SOFA score > 7

Exclusion Criteria:

* history of Diabetes mellitus
* history of hypercholesterolemia
* history of hyperhomocysteinemia
* impaired hepatic function

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Start 2006-04; Study Completion 2007-12

PRIMARY OUTCOMES:
ADMA concentration

SECONDARY OUTCOMES:
SOFA score
Organ function
Mortality

CONTACTS AND LOCATIONS:
Overall Officials: Paul am Leeuwen van, MD, PhD, Study Director — Amsterdam UMC, location VUmc
Locations (1):
- VU University Medical Center, Amsterdam, Netherlands